CLINICAL TRIAL: NCT03378921
Title: Double-blinded Randomized Placebo Controlled Study: Fecal Microbiota Transplantation in the Treatment of Chronic Pouchitis
Brief Title: Fecal Microbiota Transplantation (FMT) in the Treatment of Pouchitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Essi Karjalainen, M.D., Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HelsinkiFMT
Record Dates: First submitted 2017-12-11; First posted 2017-12-20 (Actual); Results first posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Pouchitis; Ulcerative Colitis
Keywords: FMT
MeSH Terms: conditions — Pouchitis; Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- donors feces (Experimental): Fecal microbiota transplantation (FMT) is performed by experienced endoscopists through flexible endoscopy into the afferent limb. The second FMT is installed via transanal catheter into the pouch 4 weeks after the first FMT.
  Interventions: Biological: Fecal microbiota transplantation
- patients own feces (Placebo Comparator): Fecal microbiota transplantation (FMT) is performed by experienced endoscopists through flexible endoscopy into the afferent limb. The second FMT is installed via transanal catheter into the pouch 4 weeks after the first FMT.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Fecal microbiota transplantation — Follow up of the patients include a telephone call after 12 and 26 weeks after the FMT, and a clinical control visit 52 weeks after the transplantation. The clinical part of the Pouchitis Disease Activity Index score is assessed during each call and clinical visit. Fecal stool samples for phylogenetic analysis are collected before FMT and on weeks 4, 12, 26, and 52.
  Arms: donors feces
Biological: Placebo — Follow up of the patients include a telephone call after 12 and 26 weeks after the FMT, and a clinical control visit 52 weeks after the transplantation. The clinical part of the Pouchitis Disease Activity Index score is assessed during each call and clinical visit. Fecal stool samples for phylogenetic analysis are collected before FMT and on weeks 4, 12, 26, and 52.
  Arms: patients own feces

SUMMARY:
The aim of our study is to investigate the efficacy and safety of fecal microbiota transplantation (FMT) in the treatment of antibiotic dependent chronic pouchitis. This is a double-blinded randomized placebo controlled study. 13 patients receive a fecal transplantation from the healthy tested donor and 13 patients in the control group receive their own feces.

DETAILED DESCRIPTION:
Pouchitis is the most common long term complication among patients with ulcerative colitis who have undergone restorative proctocolectomy with ileal pouch-anal anastomosis (IPAA). The etiology of pouchitis remains unclear. There is significant clinical evidence implicating bacteria in the pathogenesis. It has been shown that fecal microbiota transplantation (FMT) is an effective treatment for recurrent Clostridium difficile -infection. Case reports have also shown promising results of FMT in patients with inflammatory bowel disease. Currently there is no established effective treatment for chronic antibiotic dependent or refractory pouchitis. The aim of our study is to investigate the efficacy and safety of fecal transplantation in the treatment of chronic pouchitis instead of antibiotic therapy. Another aim is to evaluate phylogenetic analysis of the fecal microbiota trying to find microorganisms contributing to good results in fecal transplantation in IPAA patients.

Patients receive FMTs on weeks 0 and 4. Antibiotic treatment has been stopped 36 hours before the first FMT.

ELIGIBILITY:
Inclusion Criteria:

* Status post of restorative proctocolectomy with ileal pouch-anal anastomosis (IPAA) for ulcerative colitis
* Pouchitis diagnosed by the symptoms and by endoscopy including histology within 6 months prior to FMT
* Need of frequent or continuous use of antibiotics or probiotics because of the chronic pouchitis
* Availability of consecutive fecal samples during one year
* Compliance to attend FMT and control pouchoscopy after 52 weeks

Exclusion Criteria:

* Unable to provide informed consent
* Use of immunosuppressive or biological medication
* Use of corticosteroids
* Acute pouchitis
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Lepistö, PhD, MD, Study Director — Department of Gastrointestinal Surgery, Helsinki University Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

REFERENCES:
- [Derived] Karjalainen EK, Renkonen-Sinisalo L, Satokari R, Mustonen H, Ristimaki A, Arkkila P, Lepisto AH. Fecal Microbiota Transplantation in Chronic Pouchitis: A Randomized, Parallel, Double-Blinded Clinical Trial. Inflamm Bowel Dis. 2021 Oct 20;27(11):1766-1772. doi: 10.1093/ibd/izab001. PMID 33501942

RESULTS

PARTICIPANT FLOW:
Groups:
- Donors Feces: Fecal microbiota transplantation is performed by experienced endoscopists through flexible sigmoideoscopy into the afferent limb. The second FMT is installed via catheter into the pouch 4 weeks after the first FMT.
  Fecal microbiota transplantation: Follow up of the patients include a telephone call after 12 and 26 weeks after the FMT, and a clinical control visit 52 weeks after the transplantation. The clinical part of the Pouchitis Disease Activity Index score is assessed during each call and clinical visit. Fecal stool samples for phylogenetic analysis are collected before FMT and on weeks 4, 12, 26, and 52.
- Patients Own Feces: Fecal microbiota transplantation is performed by experienced endoscopists through flexible sigmoideoscopy into the afferent limb. The second FMT is installed via catheter into the pouch 4 weeks after the first FMT.
  Placebo: Follow up of the patients include a telephone call after 12 and 26 weeks after the FMT, and a clinical control visit 52 weeks after the transplantation. The clinical part of the Pouchitis Disease Activity Index score is assessed during each call and clinical visit. Fecal stool samples for phylogenetic analysis are collected before FMT and on weeks 4, 12, 26, and 52.
Period: Overall Study
Arm/Group | Donors Feces | Patients Own Feces
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donors Feces | Patients Own Feces | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (10.2) | 45.5 (11.7) | 44.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 7 | 8 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Finland | 13 | 13 | 26
Antibiotic use at time of study enrollment [Count of Participants; unit: Participants]
  continuous use | 5 | 7 | 12
  repeated | 8 | 6 | 14
Probiotics [Count of Participants; unit: Participants] | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Clinical Remission
Description: Clinical remission at week 52. All criteria need to be met: Pouchitis Disease Activity Index <7 and no need for antibiotic treatment for pouchitis during the follow up
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Donors Feces | Patients Own Feces
Number analyzed (Participants) | 13 | 13
Participants | 4 | 5
Statistical Analysis 1: Comparison: Donors Feces vs Patients Own Feces; The sample size (n = 26) was calculated according to the estimation that the remission rate in the FMT group would be 80% and 25% in the placebo group during the follow-up of 1 year. This difference of 55% was considered to be clinically meaningful. The significance level was selected to be 1%, and the power was set to 90%; Test type: Superiority; p = 0.183, Log Rank — The threshold for statistical significance was P = 0.05

2. Secondary Outcome: Evaluation of the Changes in Gut Microbiota
Description: Fecal stool samples for phylogenetic analysis are collected before FMT and on weeks 4, 12, 26, and 52.
Time Frame: 54 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Donors Feces | Patients Own Feces
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 3/13 | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donors Feces (N=13) | Patients Own Feces (N=13)
fever (General disorders) | 1 | 1
abdominal pain (Gastrointestinal disorders) | 1 | 0
fecal urgency (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT03378921/Prot_SAP_000.pdf